CLINICAL TRIAL: NCT02503748
Title: Prostate Cancer E-Health-Tutorial (PROCET): Multicenter, One-armed Intervention Study to Evaluate an Online Tutorial for Patients With Localized Prostate Cancer
Brief Title: Prostate Cancer E-Health-Tutorial
Acronym: PROCET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zurich University of Applied Sciences (Other)
Responsible Party: Principal Investigator, René Schaffert, lic.phil., Zurich University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ZH 2015-132
Record Dates: First submitted 2015-07-16; First posted 2015-07-21 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Online Tutorial
  Interventions: Other: Online tutorial

INTERVENTIONS:
Other: Online tutorial — website informing about treatment options in localized prostate cancer

SUMMARY:
In a participatory process involving urologists and former patients, the project team has developed an online information system ("tutorial") for patients with localized prostate cancer. In this field test, relevant outcomes are measured and the tutorial will be tested for its clinical applicability.

DETAILED DESCRIPTION:
Prostate cancer is the most common cancer in men: In Switzerland, every year about 6,000 men are diagnosed with prostate cancer. Men with prostate cancer at an early stage are confronted with a difficult decision: they are faced with different treatment alternatives, each with its own advantages and disadvantages. That is why a comprehensive information delivery and processing is extremely important for patients to make an informed decision.

Therefore, an online platform has been developed in collaboration with urologists and former patients. This online platform is designed to cover the individual information needs of patients with early prostate cancer. Additionally, the software aims at facilitating cooperation between patients and doctors and at increasing the satisfaction of patients with their treatment decision.

In this study, the online platform will now to be tested in clinical practice, and data will be collected for the benefit of the platform: Can the online platform actually satisfy the indivudal information needs, facilitate the therapy decision and support the cooperation between doctors and patients?

ELIGIBILITY:
Medical Inclusion Criteria:

* tumor stage: clinical stage T1 or T2
* PSA level <20 (PSA = Prostata-specific antigen)
* Gleason score <8
* age ≤ 75 years
* Assumed life expectancy ≥ 10 years

Other inclusion criteria due to the study design and the type of intervention are the following:

* patients have to be diagnosed in one of the trial sites
* Internet-enabled device in the patient's household / basal user knowledge of this device
* signing of the consent form

Exclusion Criteria:

* Impaired judgment
* Insufficient ability to read and understand German
* Emotional problems

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-07; Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
information needs (own scale) | 4 months
  questionnaire developed in line with contents of the online tutorial

SECONDARY OUTCOMES:
Decision Quality: decisional conflict (Decisional Conflict Scale) | 1 month
Decision Quality: decision regret (Decision Regret Scale) | 4 months
Role in decision making: Preferred Role (Preferred Role in Decision Making Scale) | 1 month
Role in decision making: Actual Role (Actual Role in Decision Making Scale) | 4 months
Preparation for Decision Making (Preparation for Decision Making Scale) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: René Schaffert, lic. phil., Principal Investigator — Zurich University of Applied Sciences
Locations (8):
- Switzerland (8):
  - Urologische Universitätsklinik Basel, Kantonsspital Basselland, Liestal, Basel-Landschaft
  - UrologieZentrum Bern, Bern, Canton of Bern
  - Klinik für Urologie, Luzerner Kantonsspital, Lucerne, Canton of Lucerne
  - Urologisches Kompetenzzentrum soH, Olten, Canton of Solothurn
  - Klinik für Urologie, Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Klinik für Urologie, Stadtspital Triemli, Zurich, Canton of Zurich
  - Urologie, Kantonsspital Graubünden, Chur, Kanton Graubünden
  - Urologische Klinik, Kantonsspital Münsterlingen, Münsterlingen, Thurgau